CLINICAL TRIAL: NCT01701128
Title: The Effect of Exercise Training on Gait and Quality of Life in Patients With Early Parkinson's Disease
Brief Title: The Effect of Exercise Training on Gait and Quality of Life in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol is completed
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTPD-2011
Record Dates: First submitted 2012-09-18; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Physical activity, treadmill training, rehabilitation
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Speed TT (Experimental): Walk on treadmill with progressive increases in speed
  Interventions: Other: Walking on treadmill
- Mixed TT (Experimental): Walk on treadmill with progressive increases in speed and incline
  Interventions: Other: Walking on treadmill
- Control (Active Comparator): Light-intensity exercise group, work flexibility and coordination
  Interventions: Other: Control group

INTERVENTIONS:
Other: Walking on treadmill — 3 sessions/week, 24 weeks. The heart rate does not exceed 75% of maximum heart rate (220-age) of the participant and that blood pressure does not exceed 250/115 mmHg. During the first week, the TT velocity was adjusted to 80% of preferential walking speed of the participant. The following week, the participant was encouraged to reach 90% and 100% in the third week. From the fourth week, subjects in the Speed TT had an increase in speed, depending on exercise tolerance of each participant. The TT velocity was increased by 0,2 km/h when the participant reached criteria.
  Arms: Speed TT
Other: Walking on treadmill — 3 sessions/week, 24 weeks. The heart rate does not exceed 75% of maximum heart rate (220-age) of the participant and that blood pressure does not exceed 250/115 mmHg. During the first week, the TT velocity was adjusted to 80% of preferential walking speed of the participant. The following week, the participant was encouraged to reach 90% and 100% in the third week. From the fourth week, the TT velocity was increased by 0,2 km/h or the incline of the walking surface of TT was increased by 1% alternately when the progression criteria were met.
  Arms: Mixed TT
Other: Control group — Training of the control group was characterized by light intensity exercises. For the first three months, participants performed regular exercise involving full range of motion to enhance their flexibility. For the last three months of the training programme, participants learned elements of Tai Chi and rhythmic movements of latin dance. Participants attended two 1-h supervised sessions per week and were asked to perform each week a third session at home, based on instructions in a document offered to the control group participants
  Arms: Control

SUMMARY:
The project aims to evaluate the effects of 24 weeks of treadmill training (TT), with and without a strengthening component, on functional mobility, gait and quality of life in patients with Parkinson's disease (PD). The rationale for a study of this type stems from the hypothesis that treadmill training may act as an external "pacemaker" and enhance some properties of gait. There is a need for larger scale randomized controlled trials comparing the effects of treadmill training to control groups that receive similar amounts of attention. To date, no study has combined TT and muscle strengthening, likely the optimal form of therapy. A kinesiologist supervises the training, 3 times per week, for a total of 72 one-hour exercise sessions. It is hypothesized that at the end of 6 months, treadmill training will considerably improve walking parameters and the well being of people with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease
* Stage of II or less on Hoehn and Yahr scale

Exclusion Criteria:

* Having musculoskeletal impairments or having excessive pain in any joint that could limit participation in exercise program
* Dementia (MMSE<24)
* Having balance problems
* Live beyond 45 minutes from Laval University

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in Gait speed | Baseline, 3 and 6 months
  This measure was recorded using the GAITrite system
Change in Endurance walking | Baseline, 3 and 6 months
  This measure was recorded using the 6-minutes walk test
Change in Quality of life | Baseline, 3 and 6 months
  This measure was recorded using PDQ-39

SECONDARY OUTCOMES:
Change in Postural Balance | Baseline, 3 and 6 months
  This measure was recorded using force platform PRO Balance Master®
Change in Spatiotemporal parameters of walking | Baseline, 3 and 6 months
  This measure was recorded using the GAITrite system
Change in Cognitive impairment | Baseline, 3 and 6 months
  This measure was recorded using Mini-Mental State Examination
Change in Fear of falling | Baseline, 3 and 6 months
  This measure was recorded using the ABC Scale
Change in Depression and anxiety level | Baseline, 3 and 6 months
  This measure was recorded using BDI-II
Change in Effects of symptoms and motor impairment | Baseline, 3 and 6 months
  This measure was recorded using the UPDRS

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Corbeil, Study Director — Laval University; Alexandra Nadeau, Study Director — Laval University; Emmanuelle Pourcher, Principal Investigator — Quebec Memory and Motor Skills Disorders Research Center
Locations (2):
- Canada (2):
  - Quebec Memory and Motor Skills Disorders Research Center, Québec, Quebec
  - Laval University, Québec, Quebec

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886